CLINICAL TRIAL: NCT02246309
Title: Comparison Of The Embryoscope Time-Lapse System With Standard Embryo Culture at Center for Human Reproduction(CHR):an Open Label Randomized Clinical Trial
Brief Title: Comparison Of The Embryoscope Time-Lapse System With Standard Embryo Culture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment was loaned Lifglobal, Guilford, CT, USA and had to be returned.
Sponsor: Center for Human Reproduction (Other)
Collaborators: FertiliTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ER08282014-01
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2015-12

CONDITIONS: Infertility
Keywords: Infertility; Embryo Culture; Laboratory Technique
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Embryoscope Time Lapse System (Experimental): All embryos from patients randomized to this arm will be cultured in the Embryoscope culture system from the time of insemination until the time of transfer on day 3. All staff interaction with the embryos or with maintenance or supervision of the system will be timed.
  Interventions: Device: Embryoscope Time Lapse System
- Standard Embryo Culture (Active Comparator): All embryos from patients randomized to this arm will be cultured in the standard embryo culture system from the time of insemination until the time of transfer on day 3. All staff interaction with the embryos or with maintenance or supervision of the system will be timed.
  Interventions: Device: Standard Embryo Culture

INTERVENTIONS:
Device: Embryoscope Time Lapse System — The EmbryoScope® time-lapse system is a unique platform facilitating improved IVF treatment, flexible work routines and effective communication, through comprehensive documentation of embryo development and evolving improvements in selection.
  Arms: Embryoscope Time Lapse System
Device: Standard Embryo Culture — Standard embryo culture in a Standard water jacketed carbon dioxide/low oxygen incubator system.
  Other Names: Standard water jacketed incubator system
  Arms: Standard Embryo Culture

SUMMARY:
"Embryoscopes," allow for embryo culture to be performed in an automated incubation system under time lapse photography. Manufacturers of these systems (and investigators who have used these systems) claim that the availability of 24-hour time-lapse photographic control improves embryo selection and, therefore, IVF (in vtro fertilization) pregnancy rates. They also claim that use of this system saves laboratory personnel time.

This study will randomize approximately 120 patients (60 in each arm) to standard embryo culture or to culture in an Embryoscope. The primary endpoint will be a comparison of time spent by the laboratory personnel with each system. Secondary endpoints will be IVF outcomes.

DETAILED DESCRIPTION:
A large number of IVF centers all around the world are converting from standard embryology practice, where embryos are by embryologists manually processed during culture, to so-called "embryoscopes," where embryo culture is performed in an automated incubation system under time lapse photography.

Manufacturers of these systems (and investigators who have used these systems) claim that the availability of 24-hour time-lapse photographic control improves embryo selection and, therefore, IVF pregnancy rates. They also claim that use of this system saves laboratory personnel time. The FDA has so far, therefore, approved for sale at least 2 such systems In the USA.

(i) Our analysis of the published literature has failed to find studies in support of the claim that utilization of such equipment really improves pregnancy rates with IVF; and (ii) Investigators are concerned that CHR's highly adversely selected patient population may demonstrate different utilization outcomes from standard patient populations, especially since this equipment is usually utilized to culture embryos to blastocyst stage (days 5/6), while CHR cultures most patients only to day-3.

Investigators, therefore, contacted the manufacturer of the first FDA approved system, and explained our concerns. The manufacturer agreed to loan us one of their systems for a 4-months long study free of charge (CHR just pays a nominal amount for installation and training costs) but will be financially responsible for supplies.

During these 4 months, CHR will perform an open-label prospective (registered) and randomized clinical trial, in which investigators, based on computerized randomization, will assign all CHR patients (who agree to participate with informed written consent), either to standard embryology or "embryoscope" embryology.

Recruiting approximately 30 patients per month into the study is anticipated, which would give us a population of ~n=60 in each study group.

Patient with excessive numbers of eggs retrieved (>12) will be excluded since the purpose of this study is to investigate the utility of the system in a relatively adversely selected patient population. All other patients will be offered participation.

The study will have as primary end point a time analysis of laboratory manpower, under which the time spent on each patient by embryologist will be recorded and compared and as secondary end point IVF cycle outcome, defined by number of good quality embryos available for transfer, implantation rates and clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients already planning to undergo in vitro fertilization

Exclusion Criteria:

* Patients with more than 12 oocytes will be excluded from this trial

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Barad, MD, Principal Investigator — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, New York, New York, United States

REFERENCES:
- [Result] Wu YG, Lazzaroni-Tealdi E, Wang Q, Zhang L, Barad DH, Kushnir VA, Darmon SK, Albertini DF, Gleicher N. Different effectiveness of closed embryo culture system with time-lapse imaging (EmbryoScope(TM)) in comparison to standard manual embryology in good and poor prognosis patients: a prospectively randomized pilot study. Reprod Biol Endocrinol. 2016 Aug 24;14(1):49. doi: 10.1186/s12958-016-0181-x. PMID 27553622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was completed during 3.5 months between December 2014 and March 2015, the time period our center (Center for Human Reproduction in New York City).
Pre-assignment Details: 134 patients were offered participation during the study period. Ten were excluded because they were using embryo banking. Eighty five declined participation leaving only 49 qualified and/or consented to participate.
Period: Overall Study
Arm/Group | Embryoscope Time Lapse System | Standard Embryo Culture
Started | 16 (16 patients going through Time Lapse System and 15 through Standard Embryo Culture.) | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Embryoscope Time Lapse System | Standard Embryo Culture | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (4) | 40.4 (6.97) | 39.5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Personnel Effort
Description: Number of minutes spent by laboratory personnel technical staff in support of each system
Time Frame: Three days
Measure: Mean (Standard Error); unit: technical staff minutes spent per embryo
Units Other Than Participants: embryos
Arm/Group | Embryoscope Time Lapse System | Standard Embryo Culture
Number analyzed (Participants) | 16 | 15
Number analyzed (embryos) | 44 | 42
technical staff minutes spent per embryo | 301.2 (80.8) | 137.6 (52.7)

2. Secondary Outcome: Embryo Quality
Description: Number of Grade A best quality of day 3 embryos (based on cell number and degree of fragmentation)
Time Frame: Three Days
Measure: Mean (Standard Error); unit: Embryos
Arm/Group | Embryoscope Time Lapse System | Standard Embryo Culture
Number analyzed (Participants) | 16 | 15
Embryos | 1.2 (0.3) | 1.2 (0.2)

3. Other Pre Specified Outcome: Clinical Pregnancy Rate
Description: Existence of Clinical Pregnancy documented by sonogram 4 weeks after embryo transfer
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Embryoscope Time Lapse System | Standard Embryo Culture
Number analyzed (Participants) | 16 | 15
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: One Month
Arm/Group | Embryoscope Time Lapse System | Standard Embryo Culture
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No